CLINICAL TRIAL: NCT00269347
Title: Manipulation, Exercise, and Self-Care for Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency); Berman Center for Outcomes and Clinical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP10009
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2005-12-23 (Estimated); Status verified 2005-12

CONDITIONS: Low Back Pain
Keywords: Chiropractic; Manual Therapy; Exercise; Randomized; Clinical Trial; Back Pain
MeSH Terms: conditions — Low Back Pain; Motor Activity; Back Pain | interventions — Manipulation, Chiropractic; Exercise; Self Care

INTERVENTIONS:
Procedure: Chiropractic Spinal Manipulation
Procedure: Exercise
Behavioral: Self-care

SUMMARY:
The broad, long term objective of this interdisciplinary research is to identify effective therapies for low back pain sufferers and to increase our understanding of this important condition. The primary aim is to examine the relative efficacy of chiropractic spinal manipulation, rehabilitative exercise, and self-care education in terms of patient-rated outcomes in the short and long term for non-acute low back pain.

DETAILED DESCRIPTION:
Low back pain remains an important public health problem with serious socioeconomic consequences. Despite the considerable amount of research that has been preformed, there is still a dire need for randomized clinical tiles of high methodological quality. The broad, long-term objective of this interdisciplinary research is to identify effective therapies for low back pain sufferers and increased understanding of this important condition. Building upon the principal investigators' previous collaborative research, this randomized observer-blinded clinical trial will compare the following treatment for patients with nonacute low back pain:

1. chiropractic spinal manipulation
2. rehabilitative exercise
3. self care education Theprimary aim is to examine the relative efficacy of the three interventions in terms of patient rated outcomes in the short-term (after 12 weeks) and the long-term (after 52 weeks) for nonacute low back pain.

Secondary aims include:

1. To examine the short and long-term relative cost effectiveness and cost utility of the three treatments.
2. To assess if there are clinically important differences between pre-specified subgroups of low back pain patients. Subgroups are based on duration and current episode and radiating leg pain.
3. To evaluate if there treatment group differences in objective lumbar spine function (range of motion, strength and endurance) after 12 weeks of treatment and if changes in lumbar function are associated with changes in patient rated short and long-term outcomes.
4. To identify if baseline demographic or clinical variables can predict short or long-term outcome.
5. To describe patients' interpretations and perceptions of outcome measures used in clinical trials.

ELIGIBILITY:
Inclusion Criteria: patients are 18-65 years of age; Québec task force classification 1,2,3 and 4 (this includes patients with back pain, stiffness or tenderness, with or without musculoskeletal signs and neurological signs); primary complaint of back pain, with current episode greater than or equal to six weeks duration(this includes subacute and chronic patients for whom the study treatments are an option)

-

Exclusion Criteria:

* previous lumbar spine surgery; back pain referred from local joint lesions of the lower extremities or from visceral diseases; progressive neurological deficits due to nerve root or spinal cord compression; aortic and peripheral vascular disease; existing cardiac disease requiring medical treatment; blood clotting disorders; diffuse idiopathic hyperostosis; infectious and noninfectious inflammatory or destructive tissue changes of the lumbar spine; presence of significant infectious disease, or other severe debilitating health problems; substance abuse; ongoing treatment for back pain by other health care providers; pregnant or nursing women; pain score of less than 30 percentage points; pending our current litigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-01; Study Completion 2005-04

PRIMARY OUTCOMES:
Pain (Visual Analog Scale) at baseline, weeks 4,12,26,52

SECONDARY OUTCOMES:
Disability (Modified Roland Scale) at baseline, weeks 4,12,26,52
General Health (SF-36) at baseline, weeks 4,12,26,52
Improvement (7 point scale) at baseline, weeks 4,12,26,52
Disability (NHIS) at baseline, weeks 4,12,26,52
Bothersomeness (7 point scale) at baseline, weeks 4,12,26,52
Frequency (7 point scale) at baseline, weeks 4,12,26,52
Satisfaction (5 point scale) at baseline, weeks 4,12,26,52
Depression (CES-D) at baseline, weeks 4,12,26,52
Medication use at baseline, weeks 4,12,26,52
Fear-avoidance (FABQ) at baseline, weeks 4,12,26,52
Lumbar range of motion at baseline, weeks 4,12,26,52
Lumbar strength and endurance at baseline, weeks 4,12,26,52
Health care costs and utilization at baseline, weeks 4,12,26,52

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, DC, PhD, Principal Investigator — Northwestern Health Sciences University
Locations (1):
- Northwestern Health Sciences University, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Haanstra TM, Hanson L, Evans R, van Nes FA, De Vet HC, Cuijpers P, Ostelo RW. How do low back pain patients conceptualize their expectations regarding treatment? Content analysis of interviews. Eur Spine J. 2013 Sep;22(9):1986-95. doi: 10.1007/s00586-013-2803-8. Epub 2013 May 10. PMID 23661035
- [Derived] Bronfort G, Maiers MJ, Evans RL, Schulz CA, Bracha Y, Svendsen KH, Grimm RH Jr, Owens EF Jr, Garvey TA, Transfeldt EE. Supervised exercise, spinal manipulation, and home exercise for chronic low back pain: a randomized clinical trial. Spine J. 2011 Jul;11(7):585-98. doi: 10.1016/j.spinee.2011.01.036. Epub 2011 May 31. PMID 21622028
- See also: Related Info — http://www.nwhealth.edu/research/WHCCS